CLINICAL TRIAL: NCT01060956
Title: The Clinical Impact of Isolation of Two Different Bacteria in Urinary Cultures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Shaare Zedek Medical Center, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: UTI1
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2010-02

CONDITIONS: Urinary Tract Infection
Keywords: Urinary tract infection with two bacteria in culture
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reporting on two bacteria in urine culture (Active Comparator): The microbiology laboratory will report on the isolation and susceptibilities of two different bacteria in urine culture
  Interventions: Other: reporting of two different bacteria in urine culture
- reporting "mixed growth" (Placebo Comparator): The microbiology laboratory will report on mixed growth in urine culture
  Interventions: Other: reporting "mixed growth" on urine culture

INTERVENTIONS:
Other: reporting of two different bacteria in urine culture — reporting of two different bacteria in urine culture
  Arms: Reporting on two bacteria in urine culture
Other: reporting "mixed growth" on urine culture — reporting "mixed growth" on urine culture
  Arms: reporting "mixed growth"

SUMMARY:
The purpose of this study is to determine whether identification of two different bacteria in urine culture of patients with indwelling catheter has a clinical impact - change in antibiotic, duration of antibiotic, days to clinical resolution and length of stay in hospital.

The microbiology laboratory will randomized urine cultures with two bacteria from indwelling catheter to either reporting identity and susceptibility of the bacteria or reporting "mixed growth".

ELIGIBILITY:
Inclusion Criteria:

* Adults hospitalized with indwelling urinary catheter in growth of two bacteria in urine culture

Exclusion Criteria:

* Positive blood cultures or no blood cultures taken

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Change of antibiotic treatment | During the episode of urinary tract infection

SECONDARY OUTCOMES:
Days to clinical resolution | Duration of urinary tract infection and duration of hospitalization
Increase/decrease in the spectrum of antibiotic | Duration of urinary tract infection and duration of hospitalization
Length of stay in hospital | Duration of urinary tract infection and duration of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Amos M Yinnon, MD, Prof, Principal Investigator — Hebrew university, Jerusalem, Israel